CLINICAL TRIAL: NCT01551381
Title: Double-blind, Controlled Study in Healthy and Type 2 Diabetic Subjects to Assess Safety, Tolerability and Pharmacokinetics of 28 Days EV-077 Treatment, and the Effects on Platelet Function, Vascular Inflammation and Oxidative Stress.
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of EV-077 in Type 2 Diabetic Subjects
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim review indicated that the dose selected was too high for diabetics
Sponsor: Evolva SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EV077/C005; 2011-003808-20 (EudraCT Number)
Record Dates: First submitted 2012-03-08; First posted 2012-03-12 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Type 2 Diabetes
Keywords: Safety; Tolerability; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EV-077 (Experimental): Oral administration
  Interventions: Drug: EV-077
- Placebo (Placebo Comparator): Oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EV-077 — twice daily oral administration
  Other Names: EV-077-3201-2TBS
  Arms: EV-077
Drug: Placebo — twice daily oral administration
  Arms: Placebo

SUMMARY:
The principal objective of this study is to evaluate the safety and tolerability of repeated doses of EV-077-3201-2TBS given to diabetic subjects over a 4 week treatment period. The secondary aim of this initial Phase IIa study is to evaluate the effect of multiple oral doses of EV-077-3201-2TBS on platelet function, vascular function, vascular inflammation, vascular oxidative stress, renal function and a selection of exploratory parameters and biomarkers in type 2 diabetic subjects, as well as multiple dose pharmacokinetics in diabetic subjects.

In order to ensure the safety of the diabetic subjects, initial parts of the study will evaluate the safety and tolerability of EV-077-3201-2TBS. In Part A, the safety of different doses EV-077-3201-2TBS will be investigated in healthy subjects treated for 4 weeks. In parallel, Part B will investigate potential interactions between EV-077-3201-2TBS and ASA in healthy subjects. Part C will then investigate the safety, pharmacokinetics and pharmacodynamics of EV-077-3201-2TBS in type 2 diabetic subjects with and without concomitant ASA therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 to 70 years inclusive. (NB. All females must be of non-reproductive potential, i.e. post-menopausal, post-hysterectomy, bilateral tubal ligation or bilateral oophorectomy).
* Body mass index (BMI) between 25.0 and 40.0 kg/m2 (both inclusive).
* Subjects with type 2 diabetes mellitus according to American Diabetes Association (ADA) definition for a duration of at least 3 years, on a stable therapy with oral anti-diabetic drugs (OAD) or with insulin, with or without one or two OADs or a glucagon like peptide-1 (GLP-1) agonist, or glitazones. Stable baseline therapy is defined as unchanged dose regimen for at least 3 months before administration of the study drug.
* HbA1c ≥ 6.0 and ≤ 9.0 %.
* History of hyperlipidaemia, with either elevated LDL cholesterol (>140 mg/dL) without therapy, or treatment with statins (NB. Patients on statin therapy must have a 2 week wash-out before they can enter the study).
* History of hypertension, either with systolic blood pressure levels between 140 to 160 mmHg without treatment, or treatment with ACE inhibitors or ARB, which should be stable over the previous 3 months.

Exclusion Criteria:

* Abnormal and clinically significant ECG at screening.
* Donation of any blood or plasma in the past month or in excess of 500 mL within the 12 weeks preceding screening.
* Intake of paracetamol within 7 days before start of treatment.
* Surgery or trauma with significant blood loss within the last 3 months before administration of study drug.
* Smokers (negative cotinine test required).
* Clinically significant abnormal laboratory test results during the screening as judged by the Investigator (one retest within a week is permitted, the last result being conclusive).
* Increased risk of bleeding, e.g. subjects with a history of deep cerebral bleeding or known defects of haemostasis with increased risk of bleeding, as judged by the Investigator.
* History of or presence of clinically significant diseases such as cancer, clinically significant cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, haematological, dermatological, venereal, neurological, psychiatric diseases, other major disorders as judged by the Investigator, or significant secondary diabetic complications, such as but not limited to clinically relevant peripheral neuropathy, retinopathy, diabetic foot ulcers, as judged by the Investigator.
* Supine blood pressure at screening, after resting for 5 min, of > 160 mmHg systolic or > 95 mmHg diastolic (excluding white-coat hypertension; therefore, if a repeat measurement on a second screening visit shows values within the range, the subject can be included in the trial).
* Type 1 diabetes mellitus.
* Intake of anti-inflammatory drugs except ASA (dose 75-125mg/day stable for the previous 3 months) within 14 days before start of treatment. Steroid therapy other than topical application is not allowed.
* Any treatment with diuretics (hydrochlorothiazide is allowed)
* Liver enzymes (ALT and AST) more than 1.5 times the upper limit of normal.
* Any contraindication for a therapy with ASA such as allergy to ASA, including asthma, acute gastric ulcers, haemorrhagic diathesis, renal or liver insufficiency, or heart failure.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Platelet aggregation | 8 days
  Measured at Day 8 by Multiplate® with arachidonic acid as the agonist

SECONDARY OUTCOMES:
Platelet aggregation | Days 1, 2, 8, 15, 22 and 29
  Measured at multiple time points by Multiplate (using arachidonic acid, collagen, U-46619 and ADP as agonists) and the Born method (using arachidonic acid, collagen and ADP as agonists)
Vascular inflammatory state | Baseline, 2 weeks and 4 weeks
  Changes from baseline in markers of platelet function, vascular function, vascular inflammation and vascular oxidative stress
Diabetic state | Baseline, 2 weeks and 4 weeks
  Change from baseline in fasting plasma glucose and HbA1c
Renal function | Baseline, 2 weeks and 4 weeks
  Change from baseline in urinary albumin excretion, creatinine clearance and exercise-induced microalbuminuria

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Jax, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH, Germany
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany